CLINICAL TRIAL: NCT07345026
Title: Clinical Efficacy of Acellular Dermal Matrix (Product Name: SureDerm BCS) in Breast Cancer Patients Undergoing Breast-Conserving Surgery
Brief Title: Acellular Dermal Matrix(SureDerm BCS) in Breast-Conserving Surgery for Breast Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Chang-Ik Yoon, Assistant Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XC25EIDV0042
Record Dates: First submitted 2025-09-08; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasms; Mastectomy, Segmental
Keywords: Breast Cancer; Breast-Conserving Surgery; Acellular Dermal Matrix; Oncoplastic Surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Intervention Model Description: Parallel assignment with 1:1 randomization (ADM vs no ADM)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Breast-Conserving Surgery With SureDerm (Experimental): Participants will undergo breast-conserving surgery with implantation of an acellular dermal matrix (SureDerm). All participants will also receive standard postoperative radiotherapy.
  Interventions: Device: Acellular Dermal Matrix (SureDerm BCS)
- Breast-Conserving Surgery Without SureDerm (Active Comparator): Participants will undergo standard breast-conserving surgery without the use of acellular dermal matrix. All participants will also receive standard postoperative radiotherapy.
  Interventions: Procedure: Standard Breast-Conserving Surgery

INTERVENTIONS:
Device: Acellular Dermal Matrix (SureDerm BCS) — Participants in this arm will undergo breast-conserving surgery with placement of an acellular dermal matrix (SureDerm BCS). The device is implanted during surgery to provide soft tissue support and improve cosmetic outcomes. All participants will also receive standard postoperative radiotherapy.
  Other Names: Acellular Dermal Matrix
  Arms: Breast-Conserving Surgery With SureDerm
Procedure: Standard Breast-Conserving Surgery — Participants in this arm will undergo standard breast-conserving surgery without the use of acellular dermal matrix. This procedure involves removal of the breast tumor with preservation of most of the breast tissue. All participants will also receive standard postoperative radiotherapy.
  Other Names: Lumpectomy
  Arms: Breast-Conserving Surgery Without SureDerm

SUMMARY:
The goal of this clinical trial is to evaluate whether the use of an acellular dermal matrix (SureDerm) can improve cosmetic satisfaction and is safe in women with breast cancer undergoing breast-conserving surgery.

The main questions it aims to answer are:

1. Does the use of SureDerm improve patient-reported cosmetic satisfaction after breast-conserving surgery?
2. Is the use of SureDerm safe in terms of complication rates compared to standard surgery without SureDerm?

Researchers will compare patients receiving SureDerm during surgery with patients undergoing standard breast-conserving surgery without SureDerm to see if cosmetic results and safety differ between the groups.

Participants will:

* Undergo breast-conserving surgery, with or without SureDerm (assigned randomly)
* Receive standard postoperative radiotherapy
* Complete questionnaires about cosmetic satisfaction (Breast-Q) at baseline, 1 month, and 12 months after surgery
* Be followed for complications and cosmetic assessments by physicians

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 20 to 75 years
* Diagnosed with unilateral breast cancer (ICD-10 code: C50, D05) and treated with breast-conserving surgery
* Agreed to the use of acellular dermal matrix (ADM) during surgery
* Histologically confirmed primary breast cancer
* Patients who received neoadjuvant chemotherapy are eligible
* Planned to receive standard postoperative treatment, including adjuvant radiotherapy
* Voluntarily decided to participate in the study and provided written informed consent

Exclusion Criteria:

* Evidence of distant metastasis
* Presence of infectious disease, autoimmune disease (e.g., specific rheumatologic disorders), or bleeding/coagulation disorders
* Known adverse reactions to all first-line antibiotics
* Suspected inflammatory infection of the breast prior to surgery
* Pregnant women at the time of enrollment
* Definite contraindications to the use of acellular dermal matrix
* Contraindications to radiotherapy
* Male patients
* History of another malignancy diagnosed within the past 5 years
* Patients deemed unsuitable for participation due to difficulty in data collection as judged by the investigator
* Patients unable to understand or complete the study questionnaires

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Cosmetic Satisfaction Assessed by Breast-Q | Baseline, 1 month after surgery, and 12 months after surgery
  Patient-reported cosmetic satisfaction will be assessed using the validated Breast-Q (Breast-Conserving Therapy Module) questionnaire at baseline (before surgery), 1 month after surgery, and 12 months after surgery. Scores will be reported as transformed scale scores ranging from 0 to 100, with higher scores indicating greater satisfaction. The change in scores over time will be analyzed.

SECONDARY OUTCOMES:
Incidence of Postoperative Surgical Complications after breast-conserving surgery with or without SureDerm | 1 month after surgery, and 12 months after surgery
  Complications related to breast-conserving surgery with or without SureDerm will be recorded, including wound infection, seroma, hematoma, delayed wound healing, fat necrosis, and skin necrosis. The incidence and severity of these postoperative surgical complications will be documented.
Incidence of Acellular Dermal Matrix (SureDerm)-Related Adverse Events and Local Tissue reaction | 1 month and 12 months after surgery
  Adverse events and local tissue reactions related to the use of acellular dermal matrix (SureDerm) will be assessed after surgery, including any clinically relevant local complications.
Physician-Assessed Cosmetic Outcome Using the Harvard 4-point Cosmetic Scale | 1 month and 12 months after surgery
  Cosmetic outcomes will be assessed by physicians during follow-up visits using the Harvard 4-point cosmetic scale (excellent, good, fair, poor), based on overall breast appearance, symmetry, and shape after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St. Mary's Hospital, College of Medicine, The Catholic University of Korea, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD) due to privacy concerns and regulatory restrictions. De-identified, aggregate data will be reported in peer-reviewed journals and scientific meetings.

REFERENCES:
- [Result] Gorbunov SG, Gorelov AV, Kosorotikova AI. [Etiological structure of acute respiratory viral infections in children hospitalized in 1981-1999]. Zh Mikrobiol Epidemiol Immunobiol. 2001 Nov-Dec;(6):25-7. Russian. PMID 11881489
- [Result] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246